CLINICAL TRIAL: NCT01795196
Title: The Use of Integrated Pulmonary Index (IPI) as a Determinate of Weaning Success and/or Failure in the Pediatric Population
Brief Title: Integrated Pulmonary Index (IPI) as a Determinate of Weaning Success and/or Failure in the Pediatric Population
Acronym: IPI
Status: Withdrawn | Type: Observational
Why Stopped: Lack of subjects to participate
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, David Vines, Chair and Program Director, Department of Respiratory Care, Rush University Medical Center
Other Study IDs: 10110203-IRB01
Record Dates: First submitted 2013-02-13; First posted 2013-02-20 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Respiratory Insufficiency
Keywords: pediatric extubation failure; weaning; integrated pulmonary index; mechanical ventilation; extubation readiness; respiratory monitoring tool; Endotracheal Extubation; Pediatric Intensive Care Unit; Rapid Shallow Breathing Index; Physiologic Deadspace
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Integrated pulmonary index (IPI) is a tool that monitors respiratory status. It takes into account four parameters: respiratory rate, end-tidal CO2, heart rate and O2 saturation using a pulse oximeter and specialized sidestream CO2 monitor. The device can continuously monitor and display the patient's ventilatory state as a single digit, 1-10. In addition, trends can be kept and it can provide early indication of changes in respiratory status. IPI has only been studied in pediatric patients who are under sedation; however, more uses for the monitoring tool are a possibility. One of those possibilities is to use IPI to monitor pediatric patients during the weaning and extubation process to determine if a specific number, or less than a specific number, is associated with extubation failure. Therefore, clinicians and physicians would be better able to determine if the patient is ready for extubation.

DETAILED DESCRIPTION:
This is an prospective observational study designed to collect data on the IPI in mechanically ventilated pediatric patients undergoing the weaning process and extubation using the FDA approved Capnostream 20® bedside monitor (CS20) (Covidien Inc., Mansfield, MA, USA). Inclusion criteria include patients intubated at least 24 hours who are less than 18 years of age but greater than 1 year of age. Exclusion criteria include patients less than 1 year of age or the presence of a tracheostomy tube. The IPI number will be blinded throughout the study but directly monitored values (SpO2, HR, PETCO2, RR) will be available for clinical use.

Upon meeting inclusion criteria, the subject will be given a code number to protect their identity. Study personnel will verify that the CS20 monitor matches the institutional time/date prior to use and the de-identified subject ID will be entered in the CS20 monitor. The subject will be connected to the CS20 device via a pulse oximeter probe and a CO2 sampling line attached to the ventilator circuit, both are standard of care in monitoring ventilated pediatric patients. Subjects will be monitored for 10 minutes prior to the initiation of physician directed weaning evaluation or extubation. Study personnel will verify that the IPI number on the monitor is not visible to clinicians in order to prevent changes on routine interventions.

Investigators will record date, time, and mechanical ventilator settings when the CS20 monitor is started to collect baseline data. Physician directed weaning trials or ventilator changes to test readiness for extubation will be recorded to correlate IPI values at a later date. Venous and/or arterial blood gas (ABG) data and nebulizer treatments occurring during the study will be recorded along with the PETCO2 when the ABG is drawn or nebulizer treatment administered and CS20 monitor will be marked with an event. For nebulizer treatments, mark event and also push the pump off button to pause IPI monitoring for 15 minutes in order to prevent sample line from becoming clogged. CS 20 IPI monitoring will automatically resume 15 minutes after pausing the pump. If the weaning trial is stopped or the patient is extubated, the date and time will be recorded and the monitor will be marked with an event. Subjects that fail the weaning readiness determination will have the process repeated for up to three weaning attempts. If not weaned from mechanical ventilation after the third attempt, participation in the trial will be terminated. Participation in the study will be terminated if extubation does not occur within 72 hours of enrollment.

If extubated, the event will be marked on the monitor and the date and time will be recorded on the case report form (CRF). After extubation, the subject will remain reconnected to the CS20 monitor via a PETCO2 sampling nasal cannula capable of providing supplemental oxygen and a pulse oximeter. Subjects will continue to be monitored for up to 48 hours post extubation or until transferred out of the ICU. If a subject fails extubation and requires re-intubation or use of noninvasive ventilation, the event and time will be recorded and the study will be terminated. The subject may withdraw from the study at anytime or the attending physician may terminate their participation in the trial.

Necessary protected health information (PHI) includes subject name and medical record number to track the subject at 48 hours post extubation. PHI will be maintained on a site enrollment log separate from any collected data in a locked file cabinet.

Quantitative data for this study will include the time stamped electronic parameter data by subject ID from the CS20; the CRF with de-identified demographic information, significant pulmonary medical history, ventilator parameters prior to extubation, method used to determine readiness to discontinue mechanical ventilation, number of days on mechanical ventilator, rapid shallow breathing index, VD/VT, ABG and co-morbidity, date and time of extubation and 48 hour post extubation status.

Time stamped electronic parameter data from the CS20 will be obtained from the monitor via a USB drive. Data from the CS20 will be stored in a secure computer by subject ID number. The de-identified subject demographic information, medical and pulmonary history will be obtained from the subject's electronic medical record by the study staff and recorded on the CRF. The CRFs will be stored in a Study Binder in a locked filling cabinet in the College of Sciences. The Study Binder will be stored in a secure location and the data will be retained for three years.

ELIGIBILITY:
Inclusion

* Intubated at least 24 hours
* Less than 18 years of age
* Greater than 1 year of age
* Enrollment will be stratified based upon the time a potential subject has received MV.

Exclusion

* Patients less than 1 year of age
* Presence of a tracheostomy tube

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Mechanically ventilated pediatric patients undergoing the weaning process.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
To determine if IPI predicts extubation success. | 48 hours post extubation
  The IPI number will be compared to extubation success or failure to evaluate the usefulness of the IPI as a predictor.

SECONDARY OUTCOMES:
To compare IPI to RSBI and VD/VT. | Measured prior to extubation
  To compare the rapid shallow breathing index (RSBI), physiologic dead space (VD/VT), and IPI as predictors of extubation success and / or failure in the pediatric population.
To assess is there is a correlation between PaCO2 and PetCO2. | Measured with each blood gas drawn
  The values will be measured simultaneously to assess strength of correlation. To evaluate the correlation between PaCO2 in the pediatric population.

CONTACTS AND LOCATIONS:
Overall Officials: David L Vines, MS, Principal Investigator — Chair and Program Director, Department of Respiratory Care
Locations (1):
- Rush University Medical Center- Rush Children's Hospital, Chicago, Illinois, United States